CLINICAL TRIAL: NCT06669156
Title: Insufficient Regional Anesthesia and Conversion to General Anesthesia for Cesarean Section A Qualitative Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: University Hospital of North Zealand (Unknown); Copenhagen University Hospital at Herlev (Other); Aalborg University Hospital (Other); Copenhagen University Hospital, Denmark (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, MD, PhD, Sygehus Lillebaelt
Other Study IDs: 24/67884
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section Complications; Cesarean Section Pain; Regional Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Partuients experiencing conversion of regional to general anesthesia for cesarean section: All parturients undergoing emergency or elective cesarean section in a participating hospital, who experience insufficient regional anesthesia and conversion to general anesthesia during the 1 year inclusion period

SUMMARY:
Background In Denmark, approximately 20% of all children are born via cesarean section (C-section), making it the most common surgical procedure (also internationally). The recommended anesthesia for cesarean sections is regional anesthesia (spinal or epidural, "spinal anesthesia"), as it has several advantages: the woman is awake and experiences the delivery of her child, she maintains spontaneous breathing (the risk of difficult airway management is significantly higher in pregnant women), and the risk of aspiration of stomach contents into the lungs (which is clearly increased in pregnant women) is reduced. Furthermore, regional anesthesia can contribute to early postoperative pain management to some extent.

With spinal anesthesia, most women feel pressure and touch but no pain during the cesarean section. However, some women do experience pain during the procedure, necessitating a change in the plan. If inadequate anesthesia is detected before the surgery begins, one may choose (depending on, for example, the urgency of the cesarean) to administer renewed regional anesthesia (typically an epidural). However, if the woman first experiences pain after the surgery has commenced, it is necessary to place her under general anesthesia for the remainder of the procedure. Experience shows that this process can be challenging, and there are frequent examples in clinical practice of inappropriate courses of action, where women have experienced unacceptable pain during their cesarean sections without being placed under general anesthesia. It is difficult to obtain an exact figure on how many women experience inadequate anesthesia during cesarean sections under regional anesthesia, as not all cases are recognized or followed up on. Studies indicate that up to 12% experience pain during a cesarean section.

The consequences of inadequate anesthesia for cesarean sections can be quite significant for women, including impaired bonding with the child, poorer establishment of breastfeeding, increased risk of postpartum reactions and post-traumatic stress, as well as (anecdotally) the risk of women opting out of future pregnancies, as they may be reluctant to subject themselves to a similar situation again.

Aim The aim of this study is to investigate how women experience insufficient regional anesthesia during cesarean sections that require conversion to general anesthesia. The focus is on exploring the factors that contribute positively and negatively to the woman's experience in this situation.

Method Qualitative study in six Danish hospitals.

Inclusion criteria:

* Women undergoing elective or emergency cesarean section, aged over 17 years
* Regional (spinal or epidural or combined epidural-spinal) anesthesia converted to general anesthesia intraoperatively (i.e., after surgery has commenced) due to insufficient regional anesthesia (i.e., not for obstetric indications, such as in cases of difficult fetal extraction)

Exclusion criteria:

* Does not speak Danish or English
* Does not wish to participate

The woman will be contacted for the first time on day 1 or 2 after the cesarean section (before she is discharged from the hospital). She will be informed about the project and invited to participate. As a potential project participant, she is entitled to a 24-hour consideration period, and if desired, a new contact will be arranged for the following day. If she wishes to participate, she will be contacted again after 3 months. At this time, she will receive a call to schedule a follow-up telephone interview within a few days. This will take place as a semi-structured interview, initiated with open questions and concluded with a few more specific questions. At the end of the interview, a screening for post-traumatic stress will be conducted using the PTSD-8 tool. Follow-up interviews will be recorded digitally and transcribed verbatim.

Sample Size The project encompasses all women at the participating centers who experience insufficient regional anesthesia during a cesarean section and conversion to general anesthesia during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective or emergency cesarean section, aged over 17 years
* Regional (spinal or epidural or combined epidural-spinal) anesthesia converted to general anesthesia intraoperatively (i.e., after surgery has commenced) due to insufficient regional anesthesia (i.e., not for obstetric indications, such as in cases of difficult fetal extraction)

Exclusion Criteria:

* Does not speak Danish or English
* Does not wish to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project encompasses all women at the participating centers who experience insufficient regional anesthesia during a cesarean section and conversion to general anesthesia. Based on experience, this occurs relatively infrequently, but is estimated to happen 5-10 times a year at each participating center. It is anticipated that some women may decline to participate in the project, and since cesarean sections occur at all times of the day and year, the project group may risk not identifying some cases. The number of women required to participate before a sufficient amount of information is obtained (as no new information is expected from subsequent interviews) is not known in advance; however, it is estimated that 20-30 women will need to participate. Therefore, the inclusion period is expected to last for one year.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Parturients experience of insufficient regional anesthesia and conversion to general anesthesia | Three months after the cesarean section
  Parturients experience of insufficient regional anesthesia during cesarean sections that require conversion to general anesthesia.
  Investigated through semi-structured telephone interviews.
  The focus is on exploring the factors that contribute positively and negatively to the woman's experience of this situation.

SECONDARY OUTCOMES:
Posttraumatic stress | Three months after the cesarean section
  Parturients will be screened for symptoms of posttraumatic stress, using the PTSD-8 screening tool, at the end of the follow-up telephone-interview.

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (7):
  - Viborg Hospital, Viborg, Region Midt
  - Aalborg Hospital, Aalborg
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Hillerød Hospital, Hillerød
  - Lillebaelt Hospital, Kolding, Kolding
  - Roskilde Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No